CLINICAL TRIAL: NCT05292833
Title: Study on Adherence to a Mediterranean Diet in a Population of Patients With Type 2 Diabetes Diet-Med
Brief Title: Study on Adherence to a Mediterranean Diet in a Population of Patients With Type 2 Diabetes
Acronym: DIET-MED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PHRIP 180102; 2021-A00766-35 (Other: IDRCB)
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Mediterranean Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In randomized clinical studies, the mediterranean diet has demonstrated beneficial effects on glucose and lipids levels, on body composition, on waist to hip ratio, especially in patients with type 2 diabetes. Consequently, the meditteranean diet is now recommended by experts in cardiology, nutrition and diabetology. However, many of these publications have been generated in populations living around the Mediterranean Basin. Thus, it is not sure that this diet can be used by people living outside this geographic area. We aimed to study the capacity of consecutive patients admitted in diabetology to follow the mediterranean diet recommandations during 12 months. The adherence will be studied in the real life in order to identify all limitations to follow this diet. Therefore, this study may help to find solutions to reinforce adherence to this diet.

DETAILED DESCRIPTION:
Patients older than 18 years of age and consequently admitted in the Dpt of Diabetology in the Pitié-Salpêtrière and the Georges Pompidou Euopean Hospitals will be enroled in this study. After a survey of eating habits, the 14 items of the mediterranean diet (accordingly to Schröder H et al., J Nutr 2011) will be explained. Adherence to the diet is defined by the achievement of more than 9 items from the original list of 14 items. Adhesion to the diet will be studied à 3 and 12 months by questionnaires and the analysis of olive oil consumption (urine levels of hydroxytyrosol and alpha linoleic acid levels in bloood). Consequences of adhesion to the diet on body weight, body composition, glucose and lipids levels, HbA1c and liver enzymes in blood will be collected at 3 and 12 months. At the end of the study, patients will complete a semi-quantitative questionnaire with a sociologist in order to identify main limitations to achieve items of the diet.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Patient with type 2 diabetes regardless of the hypoglycaemic treatments used and their HbA1c level.
* Patient referred to the Diabetology day hospital of the CHU Pitié-Salpêtrière and Nutrition of the HEGP for assessment of diabetes and/or for obesity assessment and dietary education as part of routine care.
* Patient accepting the constraints of the protocol after explanation of it and not opposing to participate in it.
* Patient benefiting from or entitled to health insurance coverage outside of the AME.

Exclusion Criteria:

* Patient with current or recent infections (<10 days).
* Patient with unstable neoplastic (with the exception of carcinoma in situ of the cervix or cutaneous epithelioma), hematological, psychiatric (with the exception of eating disorders (ED)).
* Pregnant or breastfeeding patient.
* Person under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with known and treated type 2 diabetes, and referred to routine care in the Diabetology Day Hospital (HDJ) of the CHU Pitié-Salpêtrière and Nutrition of the Georges Pompidou Euopean Hospital as part of a therapeutic patient education (TPE) program for education and assessment of complications.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
The percentage of patients adhering to the Mediterranean Diet | 12 months
  This pourcentage is defined as an adherence score ≥ 9 in response to the 14-item questionnaire adapted from Schröder H et al., J Nutr 2011

SECONDARY OUTCOMES:
Association between adherence and variations in the values of urinary hydroxytyrosol | at inclusion, at 3 months and at 12 months
  Questionnaire of the 14 objectives Weekly food frequency questionnaire (INPES and INVS)
Association between adherence and variations in the values of blood alpha linolenic acid | at inclusion, at 3 months and at 12 months
  Questionnaire of the 14 objectives Weekly food frequency questionnaire (INPES and INVS
Association between variations in urinary hydroxytyrosol values compared to inclusion and the declaration of an increase in olive oil consumption during follow-up. | at 3 months and 12 months
  In grams per day
Association between variations in blood alpha linolenic acid values compared to inclusion and the declaration of increased consumption of walnuts during follow-up. | at 3 and 12 months
  In grams per day
Association between variations in blood alpha linolenic acid values compared to inclusion and the declaration of increased consumption of hazelnuts during follow-up. | at 3 and 12 months
  In grams per day
Association between variations in blood alpha linolenic acid values compared to inclusion and the declaration of increased consumption of almonds during follow-up. | at 3 and 12 months
  In grams per day
To study whether adherence at baseline predicts adherence to Mediterranean Diet. | at 3 months and 12 months
  Questionnaire of the 14 objectives Weekly food frequency questionnaire (INPES and INVS)
Study whether adherence to the Mediterranean Diet modifies the frequency of food consumption | during follow-up (12 months)
  Using questionnaires from the 2011-2012 Abena study (INPES and INVS)
Describe the difficulties/barriers to the initiation of the Mediterranean Diet | at Day 15, at Day 60 and at Day 180
  By repeated telephone contacts by a dietician. During these telephone contacts, the dietician will take up the 14-item grid and evaluate with the patient the difficulties or aspects already implemented. The evolution of the 14-item grid will make it possible to analyze any difficulties encountered during contacts in order to report the progress made or the regression in the number of items made over time.
Describe the difficulties/barriers to the initiation of the Mediterranean Diet | at 12 months
  Through a validated semi-structured interview (Wycherley TP et al., Diabetic Medicine 2011) conducted by a sociologist.
  It will be a question of better understanding the experience and adherence-compliance of patients with the different elements that make up the Mediterranean Diet. The secondary objective of using this data collection tool is to understand more particularly the possible difficulties of people who are not used to consuming the foods recommended in this diet.

CONTACTS AND LOCATIONS:
Overall Officials: Céline BENOIT, Mrs, Study Director — APHP
Locations (3):
- France (3):
  - Diabetology Department - Pitié-Salpêtrière Hospital, Paris
  - Pitié Salpêtrière - Nutrition, Paris
  - Hôpital Européen Georges Pompidou - Diabétologie, Paris